CLINICAL TRIAL: NCT01178905
Title: Clinical Evaluation of a Gentle But Safe Ultrashort-term Heat Inactivation Procedure of Raw Breast Milk (BM) Containing Virulent Cytomegalovirus for Preventing CMV-infection of Preterm Infants
Brief Title: Clinical Evaluation of Ultrashort-term Heat Inactivation of Cytomegalovirus (CMV) Containing Raw Breast Milk to Prevent CMV-infection of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Prevention
Other Study IDs: BM CMV inactivation
Record Dates: First submitted 2010-07-26; First posted 2010-08-10 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-02

CONDITIONS: Cytomegalovirus Infection; Preterm Infants
Keywords: Postnatal CMV infection of preterm infants; breast milk
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mother CMV positive (Other)
  Interventions: Procedure: ultrashort heat inactivation

INTERVENTIONS:
Procedure: ultrashort heat inactivation

SUMMARY:
To evaluate, in a prospective multicenter study, ultrashort-term heat inactivation for the prevention of Cytomegalovirus (CMV) transmission in preterm infants (<32 weeks gestational age or <1500 g birth weight) under clinical conditions. Inactivation will be done only during the period of infectivity of breast milk, characterized by viral excretion strongly associated with subsequent infection, monitored by periodic virologic examinations of BM and urine of the infant. Thus the investigators hypothesis is that no CMV transmission through breast milk will occur using a gentle ultrashort heat inactivation procedure applied to infective breast milk.

The protocol has been approved by the ethics committee of Tuebingen University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* <32 Weeks or GA or <1500g BW
* mother CMV IgG positive
* breast milk feeding

Exclusion Criteria:

* parents disagree

Ages: 23 Weeks to 40 Weeks | Sex: All
Age Groups: Child
Dates: Start 2010-08; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with CMV viruria | 40 weeks gestational age, or at discharge from NICU (if this is earlier)

SECONDARY OUTCOMES:
Number of participants with specific neonatal outcome parameters as a measure of neonatal quality | 40 weeks of gestational age or at discharge from NICU (if this is earlier)
  Intracranial hemorrhage (ICH) Periventricular leucomalacia (PVL) Necrotizing enterocolitis (NEC) Bronchopulmonary dysplasia (BPD) Retinopathy of prematurity (ROP)

CONTACTS AND LOCATIONS:
Overall Officials: Rangamr Goelz, MD, Principal Investigator — Tuebingen University Hospital
Locations (1):
- Tuebingen University Hospital, Tübingen, Germany

REFERENCES:
- [Derived] Bapistella S, Hamprecht K, Thomas W, Speer CP, Dietz K, Maschmann J, Poets CF, Goelz R. Short-term Pasteurization of Breast Milk to Prevent Postnatal Cytomegalovirus Transmission in Very Preterm Infants. Clin Infect Dis. 2019 Jul 18;69(3):438-444. doi: 10.1093/cid/ciy945. PMID 30407512